CLINICAL TRIAL: NCT00631189
Title: Evaluation of the Efficacy and Safety of Rosuvastatin 5 mg Versus Pravastatin 40 mg and Atorvastatin 10 mg in Subjects With Type IIa and IIb Hypercholesterolaemia
Brief Title: Evaluation of the Efficacy and Safety of Rosuvastatin 5 mg Versus Pravastatin 40 mg and Atorvastatin 10 mg in Type IIa and IIb Hypercholesterolaemic Patients
Acronym: CAP-Chol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk / Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3560L00068; EudraCT No 2006-006697-15
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2010-09-17 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2011-06

CONDITIONS: Type IIa and IIb Hypercholesterolaemia
Keywords: dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium; Pravastatin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Rosuvastatin and Pravastatin
  Interventions: Drug: Rosuvastatin; Drug: Pravastatin
- 2 (Active Comparator): Rosuvastatin and Atorvastatin
  Interventions: Drug: Rosuvastatin; Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 5mg oral
  Other Names: Crestor
Drug: Pravastatin — 40mg oral
  Other Names: Prevachol
  Arms: 1
Drug: Atorvastatin — 10mg oral
  Other Names: Lipitor
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Rosuvastatin 5 mg as an hypercholesterolemia treatment comparatively at 2 other statins: Pravastatin 40 mg and Atorvastatin 10 mg. Treatment efficacy will be evaluated by the percentage of LDL-C variation after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* subjects presenting type IIa or IIb primary hypercholesterolaemia diagnosed for at least 3 months, in a context of primary prevention with at least two associated cardiovascular risk factors and: (i)either "naive" to all lipid-lowering therapy, (ii)or treated with a statin (treatment ongoing or stopped during the previous 8 weeks)

Exclusion Criteria:

* homozygous or heterozygous familial hypercholesterolaemia
* hypertriglyceridaemia (TG ≥ 4 g/l)
* subjects at high cardiovascular risk according to the AFSSAPS 2005 definition (coronary artery disease or history of documented vascular disease, high cardiovascular risk type 2 diabetes, subject in primary prevention with a 10-year CHD risk > 20%)
* history of adverse events or hypersensitivity to an HMG Co-A reductase inhibitor (particularly a history of myopathy)
* concomitant use of any drugs not authorized during the study
* active liver disease with elevation of serum transaminases (ASAT, ALAT) more than twice the upper limit of normal
* CPK more than 3 times the upper limit of normal
* moderate or severe renal failure (creatinine clearance < 6 ml/min)
* poorly controlled hypothyroidism; poorly controlled hypertension (DBP > 95 mm Hg and/or SBP > 180 mm Hg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Farnier, MD, Principal Investigator — Le Point Medical - Rond Point du Jour
Locations (170):
- France (170):
  - Research Site, Aix-en-Provence
  - Research Site, Allaire
  - Research Site, Amiens
  - Research Site, Ancerville
  - Research Site, Angers
  - Research Site, Annecy
  - Research Site, Anzin
  - Research Site, Arles
  - Research Site, Arthez-de-Béarn
  - Research Site, Aspach-le-Bas
  - Research Site, Aubagne
  - Research Site, Auchel
  - Research Site, Bailleul
  - Research Site, Balma
  - Research Site, Beaucaire
  - Research Site, Belfort
  - Research Site, Bersée
  - Research Site, Bézenet
  - Research Site, Béziers
  - Research Site, Biarritz
  - Research Site, Blois
  - Research Site, Bondues
  - Research Site, Bondy
  - Research Site, Bordeaux
  - Research Site, Brignoud
  - Research Site, Bruay-la-Buissière
  - Research Site, Bruges
  - Research Site, Bœrsch
  - Research Site, Cabanac-et-Villagrains
  - Research Site, Cadaujac
  - Research Site, Caen
  - Research Site, Cannes La Bocca
  - Research Site, Carnon-Plage
  - Research Site, Caylus
  - Research Site, Cernay
  - Research Site, Cestas
  - Research Site, Champcueil
  - Research Site, Chanceaux-sur-Choisille
  - Research Site, Chilly-Mazarin
  - Research Site, Clary
  - Research Site, Collioure
  - Research Site, Colombier-Fontaine
  - Research Site, Colomiers
  - Research Site, Coulonieix Chamiers
  - Research Site, Crécy-la-Chapelle
  - Research Site, Crotenay
  - Research Site, Cuise-la-Motte
  - Research Site, Derval
  - Research Site, Dijon
  - Research Site, Eckbolsheim
  - Research Site, Eckwersheim
  - Research Site, Épernay
  - Research Site, Épinal
  - Research Site, Étang-sur-Arroux
  - Research Site, Évreux
  - Research Site, Fargues-Saint-Hilaire
  - Research Site, Folembray
  - Research Site, Fos-sur-Mer
  - Research Site, Franconville
  - Research Site, Gamarde-les-Bains
  - Research Site, Gambsheim
  - Research Site, Gradignan
  - Research Site, Grand-Couronne
  - Research Site, Grendelbruch
  - Research Site, Guise
  - Research Site, Harnes
  - Research Site, Horbourg-Wihr
  - Research Site, Is-sur-Tille
  - Research Site, Ivry-sur-Seine
  - Research Site, Jarville-la-Malgrange
  - Research Site, Jeumont
  - Research Site, La Ciotat
  - Research Site, La Courneuve
  - Research Site, La Crèche
  - Research Site, La Francheville
  - Research Site, Lacrouzette
  - Research Site, Lamagistère
  - Research Site, Laval
  - Research Site, Le Bouscat
  - Research Site, Le Cannet
  - Research Site, Le Passage
  - Research Site, Les Issambres
  - Research Site, Léognan
  - Research Site, Lille
  - Research Site, Lucheux
  - Research Site, Marcq-en-Barœul
  - Research Site, Marseille
  - Research Site, Maslacq
  - Research Site, Mauguio
  - Research Site, Meaux-beauval
  - Research Site, Mennecy
  - Research Site, Mensignac
  - Research Site, Merlimont
  - Research Site, Metz
  - Research Site, Miramont-de-Guyenne
  - Research Site, Mittersheim
  - Research Site, Monfort En Chalosse
  - Research Site, Monguilhem
  - Research Site, Mont-de-Marsan
  - Research Site, Montauroux
  - Research Site, Montbéliard
  - Research Site, Monteux
  - Research Site, Montfrin
  - Research Site, Montigny-lès-Metz
  - Research Site, Montpellier
  - Research Site, Moreuil
  - Research Site, Muespach
  - Research Site, Nancy
  - Research Site, Nogent-sur-Marne
  - Research Site, Noyon
  - Research Site, Oberhausbergen
  - Research Site, Orchamps
  - Research Site, Palau-del-Vidre
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Pauillac
  - Research Site, Périgueux
  - Research Site, Pfulgriesheim
  - Research Site, Phalempin
  - Research Site, Pont-à-Mousson
  - Research Site, Pouilly-en-Auxois
  - Research Site, Poussan
  - Research Site, Pradines
  - Research Site, Puteaux
  - Research Site, Quimperlé
  - Research Site, Rognac
  - Research Site, Rohrwiller
  - Research Site, Roncq
  - Research Site, Roquevaire
  - Research Site, Roubaix
  - Research Site, Saint-Etienne
  - Research Site, Saint-Émilion
  - Research Site, Saint-Étienne-de-Montluc
  - Research Site, Saint-Girons
  - Research Site, Saint-Jean-de-Braye
  - Research Site, Saint-Leu-la-Forêt
  - Research Site, Saint-Martin-d'Oney
  - Research Site, Saint-Médard-en-Jalles
  - Research Site, Saint-Morillon
  - Research Site, Saint-Rémy
  - Research Site, Saint-Rémy-de-Provence
  - Research Site, Salles
  - Research Site, Sarlat-la-Canéda
  - Research Site, Semur-en-Auxois
  - Research Site, Serres-Castet
  - Research Site, Soissons
  - Research Site, Sorcy-Saint-Martin
  - Research Site, Strasbourg
  - Research Site, Tarare
  - Research Site, Targon
  - Research Site, Tartas
  - Research Site, Tassin-la-Demi-Lune
  - Research Site, Thônes
  - Research Site, Thun-Saint-Amand
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Trie-sur-Baïse
  - Research Site, Varces-Allières-et-Risset
  - Research Site, Vatan
  - Research Site, Vence
  - Research Site, Vélizy-Villacoublay
  - Research Site, Vieux-Boucau-les-Bains
  - Research Site, Villard-Bonnot
  - Research Site, Villette-d'Anthon
  - Research Site, Viry-Châtillon
  - Research Site, Wasselonne
  - Research Site, Wattignies
  - Research Site, Wattrelos
  - Research Site, Yerres
  - Research Site, Yffiniac

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by general practitioner. First patient included: 12 October 2007 Last patient terminated the study: 04 October 2008
Pre-assignment Details: This French multicentre, randomized double-blind study was conducted on three parallel arms. The 14-week study comprised 3 visits: a screening visit (week 0, V1), a randomization and treatment allocation visit (week 6, V2) and an evaluation visit (week 14, V3). Patients were randomized at V2 and were treated for a period of 8 weeks.
Groups:
- Initial Phase: Initial phase (between V1 and V2)
- Atorvastatin: Atorvastatin 10 mg
- Pravastatin: Pravastatin 40 mg
- Rosuvastatin: Rosuvastatin 5 mg
Period: Initial Phase
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Started | 668 | 0 | 0 | 0
Completed | 317 | 0 | 0 | 0
Not Completed | 351 | 0 | 0 | 0
Not completed — Protocol Violation | 347 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0
Period: Treatment Phase
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Started | 0 | 104 | 103 | 110
Completed | 0 | 97 | 92 | 103
Not Completed | 0 | 7 | 11 | 7
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 6 | 2
Not completed — Adverse Event | 0 | 3 | 2 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — patient did not take pravastatin | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin | Total
Number analyzed (Participants) | 0 | 104 | 103 | 110 | 317
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 57.31 (10.59) | 57.23 (10.8) | 57.04 (9.32) | 57.18 (9.95)
Gender [Number; unit: Participants]
  Female |  | 49 | 55 | 46 | 150
  Male |  | 55 | 48 | 64 | 167

OUTCOME MEASURES:

1. Primary Outcome: Change in Low Density Lipoprotein Cholesterol (LDL-C) Level After 8 Weeks
Description: To compare the percentages of LDL-C level variation. As the recruitment target was not reached at the date initially planned, and in view of the recruitment difficulties, AstraZeneca decided not to extend the patient recruitment period and to perform only a descriptive analysis of the data
Time Frame: Change from baseline and after 8 weeks of treatment
Population: 92 patients completed the study in the Pravastatin group, nevertheless, primary and secondary outcome measures are described on 91 patients in the Pravastatin arm due to one missing data in this group
Measure: Mean (Standard Deviation); unit: percentage of LDL-C decrease
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Number analyzed (Participants) | 0 | 97 | 91 | 103
percentage of LDL-C decrease |  | -39.4 (13.77) [-13.77 to 13.77] | -30.3 (15.43) [-15.43 to 15.43] | -37.6 (17.96) [-17.96 to 17.96]

2. Secondary Outcome: To Compare the Percentage of Patients Reaching the Overall LDL-C Goal According to the French Agency for the Safety of Health Products (AFSSAPS) 2005 Guidelines for the Management of Dyslipidaemic Patients
Description: Not done. As the recruitment target was not reached at the date initially planned, and in view of the recruitment difficulties, AstraZeneca decided not to extend the patient recruitment period and to perform only a descriptive analysis of the data
Time Frame: Not done
Reporting Status: Not Posted

3. Secondary Outcome: To Compare the Percentage of Patients Reaching the LDL-C Goal, in Relation to the Number of Risk Factors, According to the French Agency for the Safety of Health Products (AFSSAPS) 2005 Guidelines for the Management of Dyslipidaemic Patients
Description: as for outcome 2
Time Frame: Not done
Reporting Status: Not Posted

4. Secondary Outcome: Compare the Percentage of Total Cholesterol Variation From Baseline and After 8 Weeks of Treatment
Description: To compare the percentage of total cholesterol variation taking baseline value as a reference. As the recruitment target was not reached at the date initially planned, and in view of the recruitment difficulties, AstraZeneca decided not to extend the patient recruitment period and to perform only a descriptive analysis of the data
Time Frame: from baseline and after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: percentage of total cholesterol decrease
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Number analyzed (Participants) | 0 | 97 | 91 | 103
percentage of total cholesterol decrease |  | -28.6 (11.0) | -20.4 (11.7) | -25.2 (14.0)

5. Secondary Outcome: Compare the Percentage of HDL-C (High Density Lipoprotein Cholesterol) Variation From Baseline and After 8 Weeks of Treatment
Description: Compare the percentage of HDL-C (High Density Lipoprotein Cholesterol) variation taking baseline value as a reference and after 8 weeks of treatment. As the recruitment target was not reached at the date initially planned, and in view of the recruitment difficulties, AstraZeneca decided not to extend the patient recruitment period and to perform only a descriptive analysis of the data
Time Frame: After 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: percentage of HDL-C increase
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Number analyzed (Participants) | 0 | 97 | 91 | 103
percentage of HDL-C increase |  | 4.4 (14.3) | 7.9 (19.2) | 11.3 (20.6)

6. Secondary Outcome: Compare the Percentage of Variation From Baseline Triglycerides Values and After 8 Weeks
Description: To compare the percentage of variation from baseline triglycerides values and after 8 weeks. As the recruitment target was not reached at the date initially planned, and in view of the recruitment difficulties, AstraZeneca decided not to extend the patient recruitment period and to perform only a descriptive analysis of the data
Time Frame: Baseline and after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: percentage of triglycerides decrease
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Number analyzed (Participants) | 0 | 97 | 91 | 103
percentage of triglycerides decrease |  | -19.2 (25) | -6.1 (31.6) | -8.7 (37)

7. Secondary Outcome: Compare the Percentage of Variation From Baseline Apolipoprotein B/Apolipoprotein A1 Ratio and After 8 Weeks of Treatment
Description: To Compare the percentage of variation from baseline Apolipoprotein B/Apolipoprotein A1 ratio and after 8 weeks of treatment. As the recruitment target was not reached at the date initially planned, and in view of the recruitment difficulties, AstraZeneca decided not to extend the patient recruitment period and to perform only a descriptive analysis of the data
Time Frame: baseline and after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: percent. Apolipoprotein B/A1 decrease
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Number analyzed (Participants) | 0 | 97 | 91 | 103
percent. Apolipoprotein B/A1 decrease |  | -30.9 (14.7) | -26 (13.5) | -31.9 (17)

8. Secondary Outcome: Compare the Percentage of Variation of C-reactive Protein (CRP)
Description: To compare the percentage of variation of C-reactive protein (CRP) taking baseline values as reference. As the recruitment target was not reached at the date initially planned, and in view of the recruitment difficulties, AstraZeneca decided not to extend the patient recruitment period and to perform only a descriptive analysis of the data
Time Frame: baseline and after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: percent of variation of C-reactive prot.
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Number analyzed (Participants) | 0 | 97 | 91 | 103
percent of variation of C-reactive prot. |  | 37.3 (187.4) | 33.1 (184.2) | 15.2 (104.9)

9. Secondary Outcome: Compare the Percentage of Variation of Phospholipase A2 (PLA2)
Description: To Compare the percentage of variation of phospholipase A2 (PLA2) taking baseline value as a reference. As the recruitment target was not reached at the date initially planned, and view of the recruitment difficulties, AstraZeneca decided not to extend the patient recruitment period and to perform only a descriptive analysis of the data
Time Frame: from baseline and after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: percent of variation of phospholipase A2
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Number analyzed (Participants) | 0 | 84 | 78 | 83
percent of variation of phospholipase A2 |  | 5.6 (46.4) | 13 (73.6) | 2.9 (24.2)

10. Secondary Outcome: Compare the Numbers of Patients Achieving the LDL-C Goal According to the National Cholesterol Education Program Adult Treatment Panel III (NCEP) ATP III) Guidelines for the Management of Dyslipidaemic Patients
Description: To Compare numbers of patients achieving the LDL-C goal according to the National Cholesterol Education Program Adult Treatment Panel III (NCEP). As the recruitment target was not reached at the date initially planned, and in view of the recruitment difficulties, AstraZeneca decided not to extend the patient recruitment period and to perform only a descriptive analysis of the data. The percentage of patients achieving the NCEP-ATP III LDL-C goal. ATP III is categorized into 3 risk categories:(1) established CHD and CHD risk equivalents(2) multiple risk factors(3) zero to one (0-1) risk factor
Time Frame: from baseline and after 8 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Number analyzed (Participants) | 0 | 97 | 91 | 103
Participants |  | 42 | 22 | 38

11. Secondary Outcome: Compare the Numbers of Patients Achieving the LDL-C Goal According to the European Atherosclerosis Society (EAS) Guidelines for the Management of Dyslipidaemic Patients
Description: as for outcome 2
Reporting Status: Not Posted

12. Secondary Outcome: To Evaluate Clinical and Laboratory Safety
Description: Serious Adverse Event and Adverse Event reported throughout the study
Time Frame: duration of study
Measure: Number; unit: Adverse Events
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Number analyzed (Participants) | 317 | 97 | 92 | 103
Adverse Events | 8 | 9 | 8 | 5

ADVERSE EVENTS:
Arm/Group | Initial Phase | Atorvastatin | Pravastatin | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 2/317 | 4/97 | 1/92 | 0/103
Other Adverse Events (participants affected / at risk) | 6/317 | 5/97 | 7/92 | 5/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Phase (N=317) | Atorvastatin (N=97) | Pravastatin (N=92) | Rosuvastatin (N=103)
Coxarthrosisaggravation (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Benign prostatic nodular hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Carotid thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0
Left Lumbar Cruralgia (Nervous system disorders) | 0 | 1 | 0 | 0
VIiolent abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Worsening of gonalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Morton syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Phase (N=317) | Atorvastatin (N=97) | Pravastatin (N=92) | Rosuvastatin (N=103)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
gingival hypoplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Morton's neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
venous insufficiency (Vascular disorders) | 0 | 1 | 0 | 0
deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
knee arthroplasty joint prosthesis user (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Ear Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
lung infection (Infections and infestations) | 0 | 0 | 1 | 0
vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
As the recruitment target was not reached at the date initially planned, and in view of the recruitment difficulties, AstraZeneca decided not to extend the patient recruitment period and to perform only a descriptive analysis of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the PI wants to discuss or publish results after the trial is completed he must obtain writing authorization from AstraZeneca